CLINICAL TRIAL: NCT02545218
Title: Perineorraphy Versus Pelvic Floor Exercise - a Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Marion Ek, M.D. Ph.D., Stockholm South General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StockholmSGH
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Perineal Tear Resulting From Childbirth
Keywords: Perineum. Perineorraphy. Pelvic floor exercise.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perineorraphy. (Active Comparator): Secondary surgical repair of the perineal body. Operation is performed by a urogynecologist in an operation theater in local anesthesia. The operation aims to re-create the anatomy in the injured perineum using 2-4 sutures.
  Interventions: Procedure: Perineorraphy
- Pelvic floor exercise. (Active Comparator): Tutored pelvic floor exercise. A trained physio therapist evaluate the pelvic floor musculature and helps the patient to perform proper pelvic floor exercises using biofeedback. The patient receives a training scheme and meets the therapist regularly every second week during 4 months.
  Interventions: Other: Pelvic floor exercise

INTERVENTIONS:
Procedure: Perineorraphy — Surgery for improperly healed perineal tear
  Arms: Perineorraphy.
Other: Pelvic floor exercise — Pelvic floor exercise tutored by physio therapist.
  Arms: Pelvic floor exercise.

SUMMARY:
The perineal body is commonly injured during labor. It is possible to perform a secondary repair, a perineorraphy, which aims to reduce the symptomatology after an improperly healed perineal tear. The aim of the randomized trial is to evaluate the results of such an operation compared with conservative treatment.

DETAILED DESCRIPTION:
A randomized controlled trial which aims to evaluate objective and subjective outcomes following perineorraphy compared with pelvic floor exercise after vaginal delivery. 70 women seeking help for improperly healed perineal tear following vaginal delivery, matching our inclusion- and exclusion criteria, will be randomised into two different treatment groups, 35 to operative treatment, perineorraphy, and 35 to conservative treatment, tutored pelvic floor exercise. Assessment pre-and 6 months postoperatively will include clinical evaluation and condition specific validated questionnaires. Surgical characteristics and adverse events during follow-up are also registered.

ELIGIBILITY:
Inclusion Criteria:

* women with 2nd or 3rd degree laceration during vaginal delivery seeking for help because of troublesome symptoms from the pelvic floor
* height of perineum 2 cm or less.
* A least 6 months post partum
* stopped "exclusive breastfeeding"
* no indication for other gynecological surgical procedure

Exclusion Criteria:

* history of 4th degree laceration
* connective tissue disorder (Systemic lupus erythematosus, Sjögrens syndrome, Polymyalgia rheumatica, Marfans syndrome, Ehlers-Danlos syndrome)
* current use of systemic corticosteroids
* diabetes mellitus
* suspect occult sphincter tear on ultrasound
* history of previous urogynecological operation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Patient Global Impression of Improvement (PGI-1) | 6 months after intervention (operation or start of pelvic floor training)
  Patients own assessment of improvement 6 months after intervention using a seven grade assessment tool called PGI-1

SECONDARY OUTCOMES:
POP-Q (Pelvic organ Quantification System) | 6 months after intervention (operation or start of pelvic floor training)
  Pelvic organ prolapse is graded via the Pelvic organ Quantification System (POP-Q) into stage 0-4. It is a validated way to clinically assess and stage of the female pelvic floor.
Ultrasound of perineum | 6 months after intervention (operation or start of pelvic floor training)
  Height and depth of perineum i millimeters using ultrasonography
Pelvic floor distress inventory (PFDI 20) | 6 months after intervention (operation or start of pelvic floor training)
  20 validated questions concerning prolapse related symptoms
Pelvic Floor Impact Questionnaire (PIFQ-7) | 6 months after intervention (operation or start of pelvic floor training)
  Evaluates the effect on quality of lafe.
Prolapse Incontinence Sexual Questionnaire (PISQ) | 6 months after intervention (operation or start of pelvic floor training)
  Evaluate effects on sexual functions
Hospital Anxiety and Depression Scale (HAD) | 6 months after intervention (operation or start of pelvic floor training)
  Evaluate psychological effects
Vaginal symptoms | 6 months after intervention (operation or start of pelvic floor training)
  Three non-validated questions concerning vaginal symptoms; sensation of wideness, vaginal flatulence and excessive discharge.
Surgical complications | From surgery up to 6 months postoperatively
  Infections.Bleedings. Other complications.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Ek, M.D., Ph.D., Principal Investigator — Stockholm South General Hospital
Locations (1):
- Södersjukhuset, Stockholm, Sweden

REFERENCES:
- [Background] Woodman PJ, Graney DO. Anatomy and physiology of the female perineal body with relevance to obstetrical injury and repair. Clin Anat. 2002 Aug;15(5):321-34. doi: 10.1002/ca.10034. PMID 12203375
- [Result] Harvey MA. Pelvic floor exercises during and after pregnancy: a systematic review of their role in preventing pelvic floor dysfunction. J Obstet Gynaecol Can. 2003 Jun;25(6):487-98. doi: 10.1016/s1701-2163(16)30310-3. PMID 12806450
- [Derived] Bergman I, Westergren Soderberg M, Ek M. Perineorrhaphy Compared With Pelvic Floor Muscle Therapy in Women With Late Consequences of a Poorly Healed Second-Degree Perineal Tear: A Randomized Controlled Trial. Obstet Gynecol. 2020 Feb;135(2):341-351. doi: 10.1097/AOG.0000000000003653. PMID 31923073